CLINICAL TRIAL: NCT01113866
Title: Circulating Biomarkers as Prognostic Indicators of Death in Ambulatory Heart Failure Patients
Brief Title: Biomarkers for Prognosis of Ambulatory Chronic Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Responsible Party: Aderville Cabassi, Hypertension and Cardiorenal Disease Center Dept Internal Medicine Nephrology and Health Sciences University of Parma
Other Study IDs: CV-1997-2002_A0013-29943
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- heart failure

SUMMARY:
Biomarkers representing distinct biological domains including neurohormonal, inflammatory, metabolic-nutritional, oxidative-nitrosative and myocardial injury, might alone or in combination provide prognostic information on mortality in heart failure patients with preserved or impaired systolic function.

DETAILED DESCRIPTION:
Upon enrollment in the study, Troponin I (cTn I), BNP, norepinephrine, plasma renin activity, aldosterone, high-sensitivity C-reactive protein (hs-CRP), tumor necrosis factor-alpha (TNF-alpha), interleukin-6 (IL-6), soluble receptor of interleukin 2 (sIL-2R), leptin, prealbumin, free malondialdehyde, 15-F2t-isoprostane and protein-bound nitrotyrosine were measured in stable ambulatory, non diabetic, elderly heart failure patients. Patients were followed up until death or study termination (31st January 2009).

ELIGIBILITY:
Inclusion Criteria:

* symptomatic congestive heart failure lasting at least six months
* reduced exercise tolerance
* impaired or preserved left ventricular ejection fraction
* cardiomegaly

Exclusion Criteria:

* acute infection
* rheumatoid or other autoimmune diseases
* primary cachectic states (cancer, thyroid disease, severe liver disease)
* severe chronic lung disease
* neuromuscular disorders
* myocardial infarction within the previous 20 weeks
* diabetes mellitus
* chronic renal failure (serum creatinine level > 2.0 mg/dl, >177 micromol/L)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: heart failure patients with preserved or impaired systolic function
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 1998-10; Primary Completion 2003-05 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aderville Cabassi, MD, Principal Investigator — University of Parma
Locations (1):
- Università di Parma, Parma, Italy